CLINICAL TRIAL: NCT07383883
Title: Multimodal Tongue-Pulse Information Fusion for Syndrome Diagnosis and Cohort Study in Children With Asthma
Status: Recruiting | Type: Observational
Sponsor: Shanghai Children's Medical Center (Other)
Responsible Party: Sponsor
Other Study IDs: SCMCIRB-YJ2025013
Record Dates: First submitted 2025-12-14; First posted 2026-02-03 (Actual); Last update posted 2026-02-03 (Actual); Status verified 2026-01

CONDITIONS: Asthma
Keywords: asthma; Tongue-Pulse Diagnosis; Multimodal Phenotyping
MeSH Terms: conditions — Asthma | interventions — Observation

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- Pediatric Asthma Cohort: Children aged 5 to 18 years with a confirmed diagnosis of asthma receiving routine outpatient follow-up at Shanghai Children's Medical Center. Participants undergo non-invasive tongue image and pulse wave data collection during visits when pulmonary function testing is clinically indicated. No intervention is assigned. All clinical management follows standard care. Tongue-pulse multimodal features are analyzed in relation to asthma clinical stage, pulmonary function, airway inflammation, allergic phenotype, and asthma control status.
  Interventions: Other: No intervention (observational study)

INTERVENTIONS:
Other: No intervention (observational study) — No intervention (observational study)

SUMMARY:
Asthma is one of the most prevalent chronic respiratory diseases in children, and accurate phenotyping and disease monitoring remain challenging in routine clinical practice. This observational cohort study aims to investigate the clinical value of multimodal tongue and pulse information in the syndrome diagnosis and phenotypic characterization of pediatric asthma. Children aged 5-18 years with a confirmed diagnosis of asthma will be enrolled at Shanghai Children's Medical Center and followed in routine outpatient care.

Standardized tongue images and pulse wave data will be collected using validated acquisition devices during visits when lung function testing is performed. Quantitative features extracted from tongue and pulse data will be integrated with clinical information, including asthma stage, lung function parameters, eosinophil counts, allergic sensitization status, and Asthma Control Questionnaire-5 (ACQ-5) scores. The primary objective is to evaluate the associations between tongue-pulse multimodal features and asthma clinical stages and pulmonary function. Secondary objectives include exploring their relationships with airway inflammation and asthma control status.

This study seeks to establish a non-invasive, objective, and quantifiable approach to asthma phenotyping, providing evidence for integrating traditional diagnostic features with modern clinical data to support precision management of pediatric asthma.

DETAILED DESCRIPTION:
This study is a single-center, observational cohort study designed to investigate the clinical value of multimodal tongue and pulse characteristics in the phenotypic classification and disease monitoring of pediatric asthma. The study will be conducted at Shanghai Children's Medical Center and will enroll children aged 5-18 years with a confirmed diagnosis of asthma who are undergoing routine outpatient follow-up.

Standardized tongue images and pulse wave data will be collected using validated tongue diagnosis and pulse diagnosis devices during outpatient visits in which pulmonary function testing is clinically indicated. Tongue image acquisition will be performed under controlled lighting and positioning conditions to ensure reproducibility, while pulse wave signals will be recorded using standardized sensor placement and acquisition protocols. These procedures are non-invasive and are integrated into routine clinical workflows without altering standard medical care.

Quantitative features will be extracted from tongue images and pulse waveforms using image processing and signal analysis methods, including color space transformation, texture analysis, brightness distribution, and pulse waveform time-domain and frequency-domain parameters. These multimodal features will be systematically linked to clinical data, including asthma clinical stage (acute exacerbation, chronic persistent phase, or clinical remission), pulmonary function parameters, such as Forced Expiratory Volume in 1 second(FEV₁), Forced Expiratory Volume in 1 second/Forced Vital Capacity(FEV₁/FVC), Resistance at 5 Hz(R5), and Resistance at 20 Hz(R20), fractional exhaled nitric oxide when available, blood eosinophil counts, allergic sensitization status, and Asthma Control Questionnaire-5 (ACQ-5) scores.

The primary objective of the study is to evaluate the associations between multimodal tongue-pulse quantitative features and asthma clinical stages and pulmonary function status. Secondary objectives include exploring the relationships between tongue-pulse features and airway inflammation, asthma control level, and allergic phenotype, as well as assessing their potential utility in phenotypic stratification and longitudinal disease monitoring.

Participants will be followed according to routine clinical practice, with repeated data collection occurring only when pulmonary function testing is performed as part of standard care. Longitudinal analyses will be conducted using time-stamped clinical and tongue-pulse data to account for irregular visit intervals. This study aims to establish a non-invasive, objective, and quantifiable framework for integrating traditional diagnostic features with modern clinical indicators, providing evidence to support precision phenotyping and individualized management of pediatric asthma.

ELIGIBILITY:
Inclusion Criteria:

* Children aged 5 to 18 years.
* Clinically diagnosed asthma according to established pediatric asthma guidelines.
* Receiving routine outpatient follow-up at Shanghai Children's Medical Center.
* Able to cooperate with tongue image acquisition and pulse wave data collection.
* Able to perform pulmonary function testing when clinically indicated.
* Written informed consent obtained from parents or legal guardians, with assent from the child when appropriate.

Exclusion Criteria:

* Presence of other chronic respiratory diseases (e.g., cystic fibrosis, bronchiectasis, primary ciliary dyskinesia).
* Congenital cardiopulmonary malformations or significant cardiovascular disease.
* Acute respiratory infection or fever at the time of data collection.
* Severe systemic diseases or immunodeficiency that may affect study participation.
* Inability to comply with study procedures or incomplete clinical data.

Ages: 5 Years to 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Study Population: The study population consists of children aged 5 to 18 years with a confirmed diagnosis of asthma who are undergoing routine outpatient follow-up at Shanghai Children's Medical Center. Participants are enrolled prospectively and receive standard clinical care without any study-assigned intervention. Tongue image and pulse wave data are collected non-invasively during visits when pulmonary function testing is performed as part of routine clinical practice. Multimodal tongue-pulse features are analyzed in relation to asthma clinical stage, pulmonary function, airway inflammation, allergic phenotype, and asthma control status.
Sampling Method: Non-Probability Sample
Enrollment: 1000 (Estimated)
Dates: Start 2025-02-01 (Actual); Primary Completion 2028-01 (Estimated); Study Completion 2028-01 (Estimated)

PRIMARY OUTCOMES:
Association Between Tongue-Pulse Multimodal Features and Pulmonary Function in Pediatric Asthma | During routine outpatient visits at baseline and follow-up when pulmonary function testing is performed (up to 12 months)
  The primary outcome is the correlation between quantitative tongue-pulse multimodal features and pulmonary function parameters in children with asthma. Tongue images and pulse wave signals are collected during routine outpatient visits and analyzed to extract quantitative features, such as color, texture, and shape parameters of the tongue images, as well as pulse rate and amplitude from the pulse wave signals. Pulmonary function parameters, including FEV₁ (Forced Expiratory Volume in 1 second, measured in liters), FEV₁/FVC (Forced Expiratory Volume in 1 second to Forced Vital Capacity ratio, measured as a percentage), and airway resistance indices (R5 and R20, measured in cm H₂O/L/s), are obtained as part of standard clinical care. Correlation and regression analyses will be performed to evaluate the correlation between tongue-pulse features and pulmonary function status. Time Frame: During routine outpatient visits at baseline and follow-up when pulmonary function testing is perform

CONTACTS AND LOCATIONS:
Overall Officials: Yong Yin, Principal Investigator — Shanghai Children's Medical Center
Locations (1):
- Shanghai Children's Medical Center, Shanghai, China